CLINICAL TRIAL: NCT05921123
Title: Understanding and Anticipating Therapeutic Response And Immuno-meDIated Adverse Events in Anti-cancer Immune-checkpoint Inhibition: a Tissue Biopsy Based imaGing Study
Acronym: TADIG-R
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0219 (TADIG-R)
Record Dates: First submitted 2023-06-09; First posted 2023-06-27 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune checkpoint inhibitors (ICI) have dramatically changed the management of some types of metastatic cancer, with indications for their use continuing to expand. Despite the hope brought by these new anti-cancer molecules, the response to ICI in these poorly prognosticated cancers is heterogeneous, with a benefit observed in 20 to 30% of patients, with the combination with chemotherapy or targeted therapies offering new perspectives. By inhibiting natural checkpoints of the immune system, ICI increase the anti-tumor response, but are also responsible for immune-related adverse events (irAEs), which can be severe. There are many hypothesized mechanisms for these immune-related adverse events, but no one has ever characterized in detail the immune infiltrate within the irAEs targeted tissues.

In-depth identification of cell subpopulations within the tumor microenvironment, as well as the infiltrate within the irAEs targeted tissues, would allow the identification of new predictive factors of response and toxicity, which could be used in clinical practice at the time of diagnosis. A better understanding of immuno-mediated toxicities would allow to adapt their management, which is currently based on the inflammatory diseases they mimic. The Hyperion technology is an innovative mass cytometry imaging system, allowing the simultaneous analysis of nearly 40 markers within a tissue.

DETAILED DESCRIPTION:
Treatment by ICI opens two important fields of investigation: the first concerns the prediction of the efficacy of these treatments, an important public health issue, as they are costly and not without toxicity; and the second concerns the understanding and therefore the management of specific immuno-mediated toxicities, which may be limiting. This project will bring together several investigations, carried out by different investigators and coordinated within the B Lymphocytes, Autoimmunity and Immunotherapies (LBAI), research unit (UMR 1227) in Brest, in order to characterize the tissue actors involved in the response and the immuno-induced toxicities, in order to establish predictive factors.

1. Tissue players involved in the anti-tumour response to ICI. Predicting the response to ICI, both before the start of treatment and during the first few months, remains a real challenge, particularly in view of the possibility of pseudo-progression during the first few weeks of treatment. This question is nevertheless of vital importance, as the indications for these molecules continue to expand, with new prospects for their combination with chemotherapies or targeted therapies. The correlation between the tumour immune microenvironment and response to ICI is relatively little studied in digestive cancers, such as gastric cancer, where contradictory data exist, particularly on the prognostic value of intra-tumour lymphocytes (TILs), which may be intra-tumour or present in the stroma. Intratumoral regulatory T cells may have a negative effect on responses to ICI, in contrast to intratumoral CD8+ T cells, with a possible prognostic impact of the regulatory T cells/T cell CD8+ ratio. In contrast, the stromal infiltrate of regulatory T cells could have a positive effect. A high infiltrate of anti-tumour M2 macrophages has been associated with poorer survival in several solid cancers, in contrast to M1 macrophages in gastric cancer. In hepatocellular carcinoma, PDL1 expression by tumour cells is low and heterogeneous, but PDL1 expression by host cells, such as innate immune cells, can inhibit the cytotoxic activity of CD8+ T cells. The role of M1 macrophages remains unclear.
2. Tissue players involved in immune-mediated toxicities. By inhibiting the immune system's natural checkpoints, ICI increase the anti-tumour response, but this also leads to a loss of peripheral tolerance mechanisms and therefore to the appearance of immuno-induced side-effects (irAEs), which can affect all organs and mimic genuine autoimmune diseases. Depending on the ICI used, the type and frequency of irAEs differ, with a frequency of up to 70% for anti-PD-(L)-1 and up to 90% for anti-CTLA-4. The digestive tract is the second most frequently affected organ after the skin, with the occurrence of immuno-induced diarrhoea and colitis, sharing macroscopic features with Crohn's disease. Approximately 6% of patients may present with rheumatological involvement, with a variety of phenotypes, most often mimicking polyarthritis, polymyalgia rheumatica (PMR) or oligoarthritis of the large joints. Several hypotheses have been put forward to explain the appearance of irAEs, most of which are based on the T cell effector due to the mechanism of action of ICI. The hypothesis of cross-reactivity between a tumour antigen and a self antigen has been put forward to explain the occurrence of irAEs, as for example in cases of vitiligo occurring under immunotherapy in metastatic melanomas, with antigens shared between tumour and non-tumour melanocytes. The role of regulatory T cells (Tregs) has also been suggested. The level of circulating IL17 at the initiation of ICI has also been associated with the risk of colitis. Two recent studies have investigated synovial biopsies from immune-induced arthritis using immunohistochemistry and flow cytometry techniques after disaggregation. The first revealed the presence of memory T cells and macrophages, and demonstrated the production of TNF alpha. The other found T cells, with CD4 slightly over-represented compared with CD8, and B cells in equivalent proportion, as well as macrophages. However, no study has ever accurately characterised the inflammatory infiltrate, either within the articular synovium or within the digestive mucosa, via the simultaneous study of numerous markers, with a spatial dimension. Nor has this been done in the skin in the case of cutaneous toxicity of ICI, or in the salivary glands in the case of immuno-induced dry syndrome, for example.
3. Hyperion technology. The Hyperion imaging technology is an innovative technology within the LBAI research unit (UMR1227) in Brest, enabling the expression of 37 markers to be assessed on a tissue slide, and thus the sub-populations of immune cells within a tissue to be quantified precisely, at cellular and sub-cellular level with a resolution of 1 µm2.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old

* Treated by Immune checkpoint inhibitor (ICI) for an advanced cancer
* Treated at Brest University-Hospital, Morlaix Hospital, Quimper Hospital, Clinique Pasteur in Brest or Bordeaux University Hospital
* With a tumor or tissue biopsy (organ target of irAEs) archived in sufficient quantity for Hyperion analysis
* For the control group: patient with an inflammatory disease (autoimmune, autoinflammatory) who had a biopsy at diagnosis

Exclusion Criteria:

* Subject of guardianship (tutorship, curatorship)
* Refusal to participate
* Patient not meeting inclusion criteria for each point

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with tumors treated by immunotherapy with Immune Checkpoint Inhibitors (ICI).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-11-25 (Estimated)

PRIMARY OUTCOMES:
Tumor response according to the iRECIST criteria and occurrence of irAE over the duration of the patient's follow-up. | 24 months
  Apparition of irAE is appreciated according the physician definition. The description and grading scales of irAE found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized. A copy of the CTCAE version 5.0 can be downloaded from the CTEP web site http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm.

SECONDARY OUTCOMES:
CTCAE terminology (description of the adverse event) and grade | 24 months
  The description and grading scales of irAE found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized.
Survival (PFS et OS) | 24 months
  PFS is defined as the time from random assignment in the clinical trial to disease progression or death from any cause. OS is defined as the time from random assignment in the clinical trial to death.
Basic demographic data, disease history, nature of ICI treatment, treatment schedule | 24 months
Identification and quantification of cell subpopulations and interactions within the tumor microenvironment, differentiating ICI responders from non-responders | 24 months
Identification and quantification of cell subpopulations making up the inflammatory infiltrate in irAEs target tissues | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Brest University Hospital, Brest, France